CLINICAL TRIAL: NCT05292209
Title: ASsessment Of RiLuzole To Reduce Paroxysmal Episodes of Atrial FIbrillatiON (The SOLUTION Study)
Brief Title: RiLuzole to Reduce Atrial FIb Study Using Holter Monitoring
Acronym: SOLUTION
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Ohio State University (Other)
Responsible Party: Principal Investigator, Mark Munger, Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB_00144866
Record Dates: First submitted 2022-03-14; First posted 2022-03-23 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Atrial Fibrillation Paroxysmal
Keywords: Atrial Fibrillation Paroxysmal, Riluzole, Holter Monitoring
MeSH Terms: conditions — Atrial Fibrillation | interventions — Riluzole

STUDY DESIGN:
Intervention Model Description: A prospective, double-blind, randomized, placebo-controlled, two-arm study design in patients with PAF
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double Blind Double Dummy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active (Experimental): Riluzole 50mg BID
  Interventions: Drug: Riluzole 50 MG
- Control (Placebo Comparator): Placebo Matching Double-Dummy Pills
  Interventions: Drug: Riluzole 50 MG

INTERVENTIONS:
Drug: Riluzole 50 MG — Riluzole 50mg tablets

SUMMARY:
Atrial fibrillation (AF) is a growing clinical problem.1 AF is a highly dynamic condition involving episodes of sinus rhythm interspersed with periods of arrhythmia, becoming more difficult to terminate over time. AF carries a substantial cost, morbidity and mortality burden. There are two important approaches to the management of AF: 1). Controlling ventricular response rate without attempting to terminate or prevent AF (rate control), and 2). Attempting to control and maintain sinus rhythm (rhythm control).2 Current rhythm control with antiarrhythmic agents (AAD) is only moderately beneficial in restoration and maintenance of sinus rhythm but produce serious adverse events. AAD selection is limited based on the potential for pro-arrhythmia, patient's age, presence of structural heart disease, and renal or hepatic dysfunction. All AF anti-arrhythmic agents are associated with harm (number needed to harm 17-119).3 There remains an important need for development of an efficacious safe AAD for the control of AF. Recent published translational studies suggest that that neuronal-type Na+ channel blockade (nNav) with riluzole, a nNav inhibitor used to manage amyotrophic lateral sclerosis (ALS), can effectively suppress triggered atrial arrhythmias.4 In two independent retrospective cohorts, riluzole-treated ALS patients significantly lowered the incidence of new-onset AF. Riluzole is well-tolerated without evidence of pro-arrhythmia.5 Therefore, to assess riluzole's effects on the reduction of paroxysmal episodes of AF, we will conduct a prospective, randomized, placebo-controlled human study using holter monitors that offer continuous electrocardiographic monitoring pre- (1 month) and with exposure to riluzole or placebo (1 month) to determine statistically superior reductions in episodes of AF.

DETAILED DESCRIPTION:
HYPOTHESIS: Riluzole will statistically reduce the number of AF episodes compared to placebo over a one-month follow-up period in patients with permanent AF (PAF).

A prospective, double-blind, randomized, placebo-controlled, two-arm study design in patients with PAF will be conducted to determine efficacy by:

1. Number of episodes tachycardia in 1 month between riluzole 50mg BID versus matching placebo;
2. Time to first episode of tachycardia between riluzole 50mg BID and placebo; and
3. Safety (pro-arrhythmia, neutropenia by CBC [baseline and 1-month end] and patient signs and symptoms [weekly phone call F/U]).

SPECIFIC AIMS:

AIM 1: To determine the impact of riluzole versus placebo based on quantification of number of episodes of tachycardia between riluzole and placebo over 1 month follow-up. A second analysis of the time to first episode of tachycardia between riluzole and placebo.

AIM 2: To determine the safety of riluzole versus placebo during a 1-month administration period. Safety will be determined by appearance of pro-arrhythmia, neutropenia by CBC [baseline and 1 month end] and patient signs and symptoms [weekly phone call F/U]) compared to placebo.

Dosing of Riluzole and Placebo: Riluzole 50mg BID (at awakening and early evening) with matching placebo tablets.

STUDY DESIGN:

Double-Blind Study Protocol

The study will be conducted in accordance with the Declaration of Helsinki and have received approval from the University of Utah Institutional Review Board.

Study Population Seventy-eight adult patients with a history of symptomatic AF documented electrocardiographically within > 48 hours to 12 months will be recruited to participate in this trial. An additional 12 patients will be recruited (90 total), if necessary, for patients that are unable to complete the 30-day follow-up period. Patients will be excluded if they have a Systolic BP > 180 mmHg or Diastolic BP > 100 mmHg; atrial Fibrillation due to electrolyte imbalance, hyperthyroidism, pericarditis, or other reversible illness; NYHA FC IV Heart Failure (No ADHF Decompensation with 1 month); unstable angina, AMI, coronary surgery within 3 or coronary angioplasty within 1 month of screening; Wolff-Parkinson-White syndrome unless treated with successful ablation; infiltrative heart disease; severe valvular heart disease; history of syncope or angina precipitated by an ventricular arrhythmia, torsade de pointes, polymorphic ventricular tachycardia, or sustained monomorphic ventricular tachycardia, or cardia arrest; are prescribed VW Class I or III antiarrhythmic agents, potent CYP1A2 inhibitors; who are of child-bearing age not practicing study-defined protective measures; or are active smokers.

At screening, each patient will be have the protocol explained to them through an informed consent process, be able to ask questions, have their primary care physician / electrophysiologist review the consent form, and then make an informed decision about their participation.

For each patient that consents to participate they will have their blood drawn for a comprehensive blood chemistry-30 panel and complete blood count. If a female who is either not of childbearing potential (defined as postmenopausal for at least 1 year or surgically sterile [bilateral tubal ligation, bilateral oophorectomy, or hysterectomy]) or is practicing 1 of the following medically acceptable methods of birth control for at least one full menstrual cycle prior to screening (listed under Exclusion Criteria #13), and agrees to continue with the regimen from the time of Screening, throughout the entire study, they will be have a pregnancy test prior to initiating drug testing.

The study investigators will determine eligibility of each participant prior to randomization. If the patient is eligible to participate, a random number generated table will select study treatment: riluzole or placebo.

After each patient starts the study medication, the patient will be scheduled to undergo a cardioversion from a clinical standpoint for atrial fibrillation management. The cardioversion can be scheduled any time after the patient has been on the medication for 3 days. At the time of the cardioversion, ECG will confirm conversion to normal sinus rhythm, before the patient starts taking study medication.

During the 30-day follow-up period, heart rhythm will be monitored by continuous heart rhythm monitoring to assess AF burden. The event recorder (monitored cardiac telemetry or event monitor or holter monitor) automatically recorded atrial fibrillation based on irregularity in the R-R interval, an established method for the detection of atrial fibrillation, 6 over a period of 30 beats at any rate. Recorders will be attached to a dry-electrode (nonadhesive) belt worn around the chest (Cardiac Bio-Systems) to enable better compliance by the patients with prolonged monitoring than has been typically observed with conventional adhesive skin-contact electrodes. Patients will be instructed to wear the monitor as much as possible for 30 days. Recorded ECG data will be transmitted transtelephonically for central interpretation. All the episodes of atrial fibrillation will be adjudicated by a cardiologist who is unaware of the patient's demographic and clinical characteristics.

Throughout the 30-day study period, the patient will have access to study investigators through a 24-hour phone number to contact the study site for any reason. At day seven each patient will receive a phone call from the study site to determine return of atrial fibrillation symptoms and any study medication adverse effects.

At the end of the 30-period treatment period, each participant will return to the clinic to have their blood drawn for a comprehensive blood chemistry-30 panel and complete blood count.

Open-Label Extension Protocol

At the end of the study, all patients will become unblinded to study treatment. If the patient has no return of atrial fibrillation during the 30-day study period and is tolerating riluzole, the patient will be offered to continue treatment for an additional 90-day without charge for riluzole. During this open-label extension phase each patient will have continuous 14-day phone call follow-up by the study investigators to determine any atrial fibrillation symptoms and continued tolerance of the riluzole medication. At the end of the 90-day open-label extension period the participant will be referred to their primary physician for continued atrial fibrillation care.

STATISTICAL ANALYSIS:

Across all the analyses for the baseline characteristics, efficacy outcome and safety outcomes, p-value less than 0.05 from statistical test will be considered significant.

Baseline Characteristics Baseline characteristics of all patients in enrolled in the study will be collected. (Gender, Age, Primary Indication for Implant, CVA/TIA history, concomitant diseases/disorders, medications). Patient characteristics will be compared between the Riluzole and Placebo groups using Chi-square test and Student t-test for categorical and continuous variables, respectively.

Outcome Analysis:

Primary Efficacy Outcome - Number of tachycardia episodes per week observation. The primary outcome is the number of tachycardia episodes over treatment periods by modified intention-to-treat (at least 14 days with tachycardia data obtained). To adjust for the potential difference in the observation period attributable to any incomplete follow-up, the number of tachycardia will be divided by the seven-day interval to calculate the event density, per-patient per-week (PPPW) number of tachycardia episodes. The PPPW will be compared between the Riluzole and Placebo using a Generalized Linear Model (GLM) with a Poisson distribution and log-link function.

Secondary outcome - Time to first tachycardia event The secondary outcome of this study will be time to first tachycardia event (nth day) after the administration of either Riluzole or placebo. The cumulative proportion of patients having tachycardia by follow-up period (# days) will be calculated using Kaplan-Meier product-limit estimate where patients will be censored on the outcome date, end of 30-day follow up period, discontinuation of the assigned treatment, or loss-of-follow up for any reason including patient death. Using a Cox-proportional hazard regression model, hazard ratio for the Riluzole vs. Placebo will be calculated as a measure of treatment effect

Adverse Events. The proportion of patients reporting any adverse experience will be compared between treatment groups using Chi-square test for the two binomial probabilities. This analysis will include all patients, not just those used in the primary efficacy analysis. Adverse experiences for each patient will be reviewed. Patients who discontinued because of a noncardiac adverse experience will be recorded. Patients who discontinued because of inadequate response or continued will be recorded separately.

Statistical power and sample size. The study is aimed to determine the superiority of the Riluzole compared to the Placebo with the target incidence density ratio (primary outcome) and hazard ratio (secondary outcome) of 0.5. (Edward et al.) with α = 0.05 and β=0.8.

The minimal sample size to detect the incidence density ratio of 0.5 from a Generalized Linear Model with Poisson distribution and log-link, this study will need a total of 78 subjects. To determine the hazard ratio of 0.5 with the overall event rate of 50% assuming that a third of the riluzole and two-third of the placebo group have at least one tachycardia during the follow-up, the total sample size must be greater than or equal to 104. Thus 55 patients randomly allocated to each group will be sufficiently powered and allows nominal attrition (<> 5%). Sample size estimation was performed using STATA 13.0 (College Station, TX: StataCorp LP).

ELIGIBILITY:
Inclusion Criteria:

* Males or Female adult patients (> 18 years old) with a history of symptomatic AF documented electrocardiographically within > 48 hours to 12 months before enrollment.
* Is able to provide written informed consent to participate in the study and is able to understand the procedures and study requirements.
* Must voluntarily sign and date an informed consent form that approved by the University of Utah IRB before the conduct of any study-specific procedure.
* Will be anti-coagulated or is already anti-coagulated for planned cardioversion.
* Is planned to undergo a cardioversion.
* Patients who are not being treated with an anti-arrhythmic agent per their physician's treatment plan

Exclusion Criteria:

* Systolic BP > 180 mmHg or Diastolic BP > 100 mmHg;
* Atrial Fibrillation due to electrolyte imbalance, hyperthyroidism, pericarditis, or other reversible illness;
* NYHA FC IV Heart Failure (No ADHF Decompensation with 1 month);
* Unstable Angina, AMI, coronary surgery within 3 or coronary angioplasty within 1 month of screening;
* Wolff-Parkinson-White syndrome unless treated with successful ablation;
* Infiltrative heart disease;
* Severe valvular heart disease;
* History of syncope or angina precipitated by an ventricular arrhythmia;
* History of torsade de pointes;
* Any polymorphic ventricular tachycardia;
* Sustained monomorphic ventricular tachycardia, or cardia arrest;
* Class I or III antiarrhythmic agents;
* Females of childbearing age. If female, is either not of childbearing potential (defined as postmenopausal for at least 1 year or surgically sterile [bilateral tubal ligation, bilateral oophorectomy, or hysterectomy]) or is practicing 1 of the following medically acceptable methods of birth control for at least one full menstrual cycle prior to screening (see below), and agrees to continue with the regimen from the time of screening, throughout the entire study they are excluded;
* Hormonal methods such as oral, implantable, injectable, vaginal ring, or transdermal contraceptives for a minimum of 3 full cycles (based on the subject's usual menstrual cycle period) before study medication administration
* Total abstinence from sexual intercourse since the last menses before study medication administration
* Intrauterine device
* Double-barrier method (condoms, sponge, or diaphragm with spermicidal jellies or cream);
* Aminotransferases > 5 x ULN (Test in the last 3 months);
* CYP 1A2 Potent Inhibitors including cimetidine, ciprofloxacin, enoxacin, rifampin, barbiturates, and fluvoxamine; and
* Active tobacco use. (i.e., smoking)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2022-06-15 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Episodes of Tachycardia | 30 Days
  Number of episodes of atrial fibrillation in 1 month between riluzole 50mg BID versus matching placebo;
Time to First Tachycardia Episode | 30 Days
  Time to first episode of atrial fibrillation between riluzole 50mg BID and placebo

SECONDARY OUTCOMES:
Safety of Riluzole Pro-Arrhythmia | 30 Days
  1. Pro-arrhythmia measured as number of episodes of V tachycardia over 30 days
Safety of Riluzole Neutropenia | 30 days
  Neutropenia measured by change on CBC [baseline and 1-month end] and patient signs and symptoms [weekly phone call F/U]).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD Sharing Plan: with Dr. Radwanski at the Ohio State University. The study protocol, statistical analysis plan, and clinical study report (only deidentified data) will be shared.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Within 30 days after completion of last patient
Access Criteria: De-identified data only